CLINICAL TRIAL: NCT03783312
Title: Effects of Preemptive Intravenous Paracetamol and Ibuprofen on Headache and Myalgia in Patients After Electroconvulsive Therapy
Brief Title: Effects of Preemptive Paracetamol and Ibuprofen on Headache and Myalgia in Patients After Electroconvulsive Therapy
Acronym: ECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Erol Karaaslan, Asst. Prof. Dr. Erol Karaaslan, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ekaraaslan1
Record Dates: First submitted 2018-12-14; First posted 2018-12-21 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain; Myalgia; Headache
Keywords: Electroconvulsive therapy; Intravenous paracetamol; Intravenous ibuprofen; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Myalgia; Headache | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Placebo-Controlled Clinical Trial
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): 250 ml saline will be administered 60 minutes before the onset of Electroconvulsive therapy procedure. Electroconvulsive therapy (ECT) is one of the effective and life-saving treatment modality used in psychiatry for a long time because it responds more rapidly than pharmacological treatment.
  Interventions: Drug: placebo
- paracetamol (Active Comparator): 1 g paracetamol will be administered 60 minutes before the onset of Electroconvulsive therapy procedure. Electroconvulsive therapy (ECT) is one of the effective and life-saving treatment modality used in psychiatry for a long time because it responds more rapidly than pharmacological treatment.
  Interventions: Drug: paracetamol
- ibuprofen (Active Comparator): 800 mg ibuprofen will be administered 60 minutes before the onset of Electroconvulsive therapy procedure. Electroconvulsive therapy (ECT) is one of the effective and life-saving treatment modality used in psychiatry for a long time because it responds more rapidly than pharmacological treatment.
  Interventions: Drug: ibuprofen

INTERVENTIONS:
Drug: placebo — 250 ml saline will be administered 60 minutes before the onset of Electroconvulsive therapy procedure. All administrations will be applied through IV infusion over 60 minutes.
  Arms: placebo
Drug: paracetamol — 1 g paracetamol will be administered 60 minutes before the onset of Electroconvulsive therapy procedure. All administrations will be applied through IV infusion over 60 minutes.
  Arms: paracetamol
Drug: ibuprofen — 800 mg ibuprofen will be administered 60 minutes before the onset of Electroconvulsive therapy procedure. All administrations will be applied through IV infusion over 60 minutes.
  Arms: ibuprofen

SUMMARY:
The primary aim this prospective, randomized, double-blind, placebo-controlled clinical trial is to compare the analgesic effects of preemptive intravenous paracetamol and ibuprofen on headache and myalgia, and secondary aim is to evaluate the effects on hemodynamics, duration of seizure and postoperative side effects in patients who underwent electroconvulsive therapy .

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is one of the effective and life-saving treatment modality used in psychiatry for a long time because it responds more rapidly than pharmacological treatment. ECT is used safely in treatment-resistant depression, and in psychiatric disorders such as mania, schizoaffective disorder, schizophrenia, catatonia, and neuroleptic malignant syndrome. Treatment response to ECT in patients with severe depression and mania was reported as 83% and 78%, respectively.

The electrical stimulation applied to the brain in ECT stimulates neuronal cells and a generalized tonic clonic seizure usually occurs for 20 to 60 seconds. ECT is performed 3 times a week for a total of 6-12 sessions.

The exact mechanism of ECT is not known, but (1) release of neurotransmitters such as dopamine, serotonin and norepinephrine (2) hypothalamic release of hormones such as prolactin and endorphins (3) gamma-aminobutyric acid conduction (4) increase in neurotrophic signaling and neurogenesis induction, and (5) factors such as changing the connection between different parts of the brain are thought to play a role.

Although studies have shown the effectiveness of ECT in treatment, low mortality and morbidity rates, and several side effects have been reported. These; oral cavity damage to tongue, teeth, implants or intraosseous denture supports; confusion; dizziness; nausea and vomiting; headache, and myalgia.

The etiology of headache after ECT is not fully understood; however, studies suggest that rapid contraction of the temporalis and masseter muscles due to ECT, vascular changes and serotonergic neurotransmission trigger headache. Headaches have been reported to be mild, moderate or severe and, in some cases, resistant to treatment.

One of the most common side effects of ECT is myalgia. In some cases it is quite severe. The mechanism of myalgia is not fully known. Muscle contractions and muscle fasciculation due to succinylcholine use are thought to be effective in the formation of myalgia during the seizure induced by ECT. There are also studies showing that the using of succinylcholine is effective on the severity of myalgia.

In cases with myalgia and headache are severe and untreated, patients cannot tolerate the pain. This may lead to discontinuation of treatment. Effective analgesic treatment is important for continued treatment and patient comfort.

Painful stimuli from damaged tissue causes sensitization in peripheral and central pain pathways. Preemptive analgesia is a treatment that was initiated before the surgical procedure to reduce this sensitization and to inhibit the response to nociceptive stimuli. Preemptive analgesia has been described as an effective method to prevent headache after ECT.

The primary aim this prospective, randomized, double-blind, placebo-controlled clinical trial is to compare the analgesic effects of preemptive intravenous paracetamol and ibuprofen on headache and myalgia, and secondary aim is to evaluate the effects on hemodynamics, duration of seizure and postoperative side effects in patients who underwent ECT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with major depression
* Patients with American Society of Anesthesiologists (ASA) scores I or II
* Between 18-65

Exclusion Criteria:

* Patients with ASA scores III/IV,
* Under the age of 18,
* Over the age of 65,
* Myocardial infarction,
* Congestive heart failure,
* Pulmonary disease,
* Stroke history,
* Bleeding disorder,
* Hepatic and renal dysfunction,
* Pregnant,
* Migraine history,
* Allergy of nonsteroidal anti-inflammatory drugs, paracetamol, propofol,
* Neuromuscular disease,
* Peptic ulcer disease,
* Intracranial hypertension,
* Glaucoma
* Patients who did not give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | From end of anesthesia (15 minutes after anesthesia) to after 24 hours, up to 24 hours
  Visual Analog Scale (Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.It is often used in epidemiologic and clinical research to measure the intensity or frequency of various pain. minimum: 0, maximum: 10, 0: no pain, 1-3: mild pain, 4-6: moderate pain, 7-10: severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Karaaslan, Asst Prof, Study Director — Inonu University Medical Faculty
Locations (1):
- Erol Karaaslan, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinwiddie SH, Huo D, Gottlieb O. The course of myalgia and headache after electroconvulsive therapy. J ECT. 2010 Jun;26(2):116-20. doi: 10.1097/YCT.0b013e3181b07c0a. PMID 19710619

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03783312/Prot_SAP_000.pdf